CLINICAL TRIAL: NCT02249013
Title: Short-course Hyperthermic IntraPEritoneal Chemotherapy (HIPEC) at Interval Debulking Surgery for High Tumor Burden Ovarian Cancer
Brief Title: Short-course HIPEC in Advanced Epithelial Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Professor Fernando Figueira Integral Medicine Institute (Other)
Collaborators: Hospital de Câncer de Pernambuco (Recife/PE) (Unknown); AC Camargo Cancer Center (São Paulo/SP) (Unknown); Instituto Brasileiro de Controle do Câncer (São Paulo/SP) (Unknown); Hospital de Cancer de Barretos - Fundacao Pio XII (Barretos/SP) (Unknown); Hospital Sao Jose (Criciuma/SC) (Unknown); Hospital de Base do Distrito Federal (Brasilia/DF) (Unknown)
Responsible Party: Principal Investigator, Thales Paulo Batista, Consultant Physician and Researcher, Professor Fernando Figueira Integral Medicine Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U1111-1158-0472; 18388113.4.0000.5201 (Other: CAAE)
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Ovarian Cancer
Keywords: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Cytoreduction Surgical Procedures; Hyperthermic Intraperitoneal Chemotherapy; Neoadjuvant Therapy; Carboplatin; Paclitaxel; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HIPEC (Experimental): Neoadjuvant Chemotherapy (NACT) followed by Cytoreductive Surgery (CRS) under a Fast-track recovery strategy plus Hyperthermic Intraperitoneal Chemotherapy (HIPEC) and thus, Adjuvant Chemotherapy
  Interventions: Procedure: Cytoreductive Surgery (CRS); Procedure: Hyperthermic Intraperitoneal Chemotherapy (HIPEC); Drug: Neoadjuvant Chemotherapy (NACT); Drug: Adjuvant Chemotherapy; Procedure: Fast-track recovery strategy

INTERVENTIONS:
Procedure: Cytoreductive Surgery (CRS) — CRS was performed with standard peritonectomy procedures and visceral resections directed towards complete elimination of tumors from the abdominopelvic cavity.
Procedure: Hyperthermic Intraperitoneal Chemotherapy (HIPEC) — HIPEC was performed according to the closed-abdomen technique using CDDP (25 mg/L of perfusate/m2, total limit of 240mg) for the first 10 patients and thus, using CDDP plus Doxorubicin (15mg/L) thereafter, both for 30 minutes, with an intra-abdominal target temperature of 41-43°C. Perfusate (2L/m2, ranging from 4L to 6L) was circulated using an extracorporeal circulation device (Performer HT; RAND, Medolla, Italy) at a flow rate of 700 ml/min.
Drug: Neoadjuvant Chemotherapy (NACT) — Systemic chemotherapy included the standard combination of carboplatin (AUC 6) and paclitaxel (175 mg/m2) administered every 21 days as neoadjuvant (2-4 cycles) plus adjuvant regimens (2-4 cycles), in the total of 6 cycles of systemic chemotherapy.
  Other Names: Carboplatin; Paclitaxel
Drug: Adjuvant Chemotherapy — Systemic chemotherapy included the standard combination of carboplatin (AUC 6) and paclitaxel (175 mg/m2) administered every 21 days as neoadjuvant (2-4 cycles) plus adjuvant regimens (2-4 cycles), in the total of 6 cycles of systemic chemotherapy.
  Other Names: Carboplatin; Paclitaxel
Procedure: Fast-track recovery strategy — A comprehensive fast-track program was applied to accelerate recovery, reduce morbidity, and shorten convalescence for patients enrolled in our trial.

SUMMARY:
This is an open-label, multicenter, single-arm, feasibility phase 2 trial on safety and efficacy of short-course regimen of intra-operative Hyperthermic Intraperitoneal Chemotherapy (HIPEC) at the time of fast-track interval debulking surgery (IDS) following neoadjuvant chemotherapy (NACT) for high tumor burden epithelial ovarian cancer (EOC).

DETAILED DESCRIPTION:
This study was initially designed to explore the safety and efficacy of short-course HIPEC in terms of median progression-free survival (PFS) as the primary outcome. However, due to slow accrual, the design was subsequently amended to explore the primary outcome measure of PD9 (i.e.: proportion of patients with disease progression or death occurring within 9 months of IDS plus HIPEC). The hypothesis was the short-course HIPEC could decrease PD9 with low rates of morbidity and mortality. In these settings, we explore a comprehensive treatment approach involving fast-track advanced cytoreductive surgery (CRS) plus short-course HIPEC at the time of IDS following NACT for high tumor burden patients with stage III-IV ovarian cancer. Advanced CRS was performed with standard peritonectomy procedures and visceral resections directed towards complete elimination of tumors from the abdominopelvic cavity, and fast-track recovery strategies were also applied to improve patient outcomes. HIPEC was performed according to the closed-abdomen technique using CDDP (25 mg/L of perfusate/m2, total limit of 240mg) or CDDP plus Doxorubicin (15mg/L) for 30 minutes, with an intra-abdominal target temperature of 41-43°C. Perfusate (2L/m2, ranging from 4L to 6L) was circulated using an extracorporeal circulation device (Performer HT; RAND, Medolla, Italy) at a flow rate of 700 ml/min. Systemic chemotherapy included the standard combination of carboplatin and paclitaxel as neo-adjuvant plus adjuvant regimens.

ELIGIBILITY:
* Inclusion Criteria:

  * Patients with no previous treatment and candidates for elective surgery with histological diagnosis of epithelial ovarian carcinoma;
  * Clinical stage IIIB to IV, without suspicion of extra-abdominal metastasis;
  * No other malignancies in activity;
  * No previous treatments such as radiation, chemotherapy (except neoadjuvant chemotherapy in the study protocol) or major abdominal surgery;
  * Absence of neuro-psychiatric disorders, history of drug allergies, and pregnancy or breast feeding;
  * Aged between 18 and 70 years;
  * Performance status 0-2 (ECOG, Eastern Cooperative Oncology Group) and / or greater than 70 points by the Karnofsky scale;
  * Appropriated cardio-respiratory, hepato-renal and hematological reserves;
  * Signing of the Consent Form.
* Exclusion Criteria:

  * Evidence of extensive retroperitoneal lymph node involvement or unresectable disease (i.e., massive involvement of the small bowel, mesentery, or hepatic pedicle, and ureteral or biliary obstruction) at the time of CRS/HIPEC;
  * Residual disease after the CRS greater than or equal to 2.5 mm (CC-2 and CC-3);
  * Limiting obesity for CRS or HIPEC;
  * Disease progression, apparent or confirmed uncontrolled infection, or health impairment during NACT.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2021-02-23 (Actual); Study Completion 2021-02-23 (Actual)

PRIMARY OUTCOMES:
PD9 | 9 months
  Proportion of patients with disease progression or death occurring within 9 months of IDS plus HIPEC

SECONDARY OUTCOMES:
Postoperative 30-day mortality rate | 30 days
  Mortality rates up to 30-day after surgery
Postoperative complication rates | 30 days
  Complications rates up to 30-day after surgery
Assessment of quality of life (QLQ-C30/EORTC) | Baseline (i.e., at the time of hospital admission for IDS plus HIPEC); after CRS/HIPEC (i.e., at the time of restarting the systemic chemotherapy); after protocol (i.e., at 3-6 weeks after the last syst
  Assessment of quality of life according to the QLQ-C30/EORTC scales.
Overall survival (OS) | 24 months
  We defined OS as the time from starting the NACT to death.
Progression-free Survival (PFS) | 24 months
  We defined PFS as the time from starting the NACT to disease progression.
Disease-free Survival (DFS) | 24 months
  We defined DFS for patients without no gross residual disease as the time from IDS plus HIPEC to disease progression.

OTHER OUTCOMES:
Time to start chemotherapy after surgery | An expected range of 4 to 8 weeks
  Time to start adjuvant chemotherapy after surgery (CRS).
Length of ICU and hospital stay | An expected range of 5 to 30 days
  Length of ICU and hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Thales P Batista, MD, MS, Principal Investigator — Professor Fernando Figueira Integral Medicine Institute

IPD SHARING:
Plan to Share IPD: No
We have no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Result] Batista TP, Carneiro VCG, Tancredi R, Teles ALB, Badiglian-Filho L, Leao CS. Neoadjuvant chemotherapy followed by fast-track cytoreductive surgery plus short-course hyperthermic intraperitoneal chemotherapy (HIPEC) in advanced ovarian cancer: preliminary results of a promising all-in-one approach. Cancer Manag Res. 2017 Dec 13;9:869-878. doi: 10.2147/CMAR.S153327. eCollection 2017. PMID 29263704
- [Result] Batista TP, Badiglian Filho L, Leao CS. Exploring flow rate selection in HIPEC procedures. Rev Col Bras Cir. 2016 Dec;43(6):476-479. doi: 10.1590/0100-69912016006014. English, Portuguese. PMID 28273222
- [Result] Lustosa RJC, Batista TP, Carneiro VCG, Badiglian-Filho L, Costa RLR, Lopes A, Sarmento BJQ, Lima JTO, Mello MJG, LeAo CS. Quality of life in a phase 2 trial of short-course hyperthermic intraperitoneal chemotherapy (HIPEC) at interval debulking surgery for high tumor burden ovarian cancer. Rev Col Bras Cir. 2020;47:e20202534. doi: 10.1590/0100-6991e-20202534. Epub 2020 Jul 10. English, Portuguese. PMID 32667582
- See also: The first paper describing early outcomes and insights after an interim analysis of our pioneering clinical trial in Brazil — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5732565/
- See also: A technical note exploring the dynamic relationships between flow rates and temperature parameters in the first cases of our study. — http://www.scielo.br/scielo.php?script=sci_arttext&pid=S0100-69912016000600476&lng=en&nrm=iso&tlng=en